CLINICAL TRIAL: NCT04192201
Title: A Real-world Study for Patients With Multiple Pulmonary Ground-glass Nodules
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Tongji Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: TJ-LC-02
Record Dates: First submitted 2019-09-23; First posted 2019-12-10 (Actual); Last update posted 2019-12-10 (Actual); Status verified 2019-10

CONDITIONS: Multiple Pulmonary Nodules
Keywords: Multiple Pulmonary Nodules; Lung Neoplasms
MeSH Terms: conditions — Multiple Pulmonary Nodules; Lung Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood or tissues of Multiple Pulmonary Nodules in a patient.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The purpose of this study is to actively monitor patients with multiple pulmonary Ground-glass Nodules (GGNs), in order to provide evidence for multiple GGNs treatment.

DETAILED DESCRIPTION:
Multiple pulmonary GGNs are very commonly identified particularly as increasing numbers of CT scans are performed as part of routine lung cancer screening. At the same time, the ideal solution for these cases continues to be debated. This aim of this study is to learn more about the effects of multiple factors on outcome of multiple pulmonary GGNs, such as patients' clinical characteristics, CT features and different pathological types. Furthermore, the optimal timing of surgery and the effect of different surgical choices on the prognosis of patients with multiple GGNs will be investigated.

ELIGIBILITY:
Inclusion Criteria:

1. Age greater than 18 years
2. Have two or more GGNs on CT imaging
3. Diameter of GGNs > 5mm and ≤ 3cm
4. GGNs must be greater than half ground glass

Exclusion Criteria:

1. patients who have a history of lung cancer
2. patients who have undergone chemotherapy, radiotherapy or targeted therapy before surgery
3. pregnant women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who were diagnosed with multiple GGNs by chest CT scan in a hospital.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2019-12-31 (Estimated); Primary Completion 2021-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
5-year overall survival [Time Frame: From date of the recruitment, assessed up to 60 months] | October 31, 2024
  5-year overall survival

SECONDARY OUTCOMES:
5-year Progression-Free-Survival [Time Frame: From date of the recruitment, assessed up to 60 months] | October 31, 2024
  5-year Progression-Free-Survival
Recurrence-free survival [Time Frame: From date of the recruitment, assessed up to 60 months] | October 31, 2024
  Recurrence-free survival

CONTACTS AND LOCATIONS:
Locations (1):
- Tongji Hospital, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: Undecided